CLINICAL TRIAL: NCT06649253
Title: REALL CD9 : Molecular Mechanisms Involved in Relapses of Childhood B-acute Lymphoblastic Leukaemia, Role of Non-coding RNA in CD9 Gene Regulation
Brief Title: Childhood B-acute Lymphoblastic Leukaemia and Role of CD9 Gene Regulation in Relapse
Acronym: REALL CD9
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC23_8885_REALLCD9
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Lymphoblastic, Acute, Pediatric
Keywords: CD9; miRNA; gene regulation
MeSH Terms: conditions — Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): All included patients. Bone and blood sampling
  Interventions: Other: Sampling bone tissue and blood

INTERVENTIONS:
Other: Sampling bone tissue and blood — Extra tube collection of bone and blood will be collected during routine care sampling interventions at the diagnosis, after the first phase of treatment and after relapse, if it occurs.

SUMMARY:
B-acute lymphoblastic leukaemia (B-ALL) is the most common cancer in children, with 20% of patients relapsing. CD9, a transmembrane protein, is linked to the migratory and adhesion capacities of leukaemia cells and could be associated with relapses. The aim of this project is to understand how CD9 regulation can be a marker of potential relapses, using bone and blood sampling of newly diagnosed patients at 3 crucial moments of therapy.

DETAILED DESCRIPTION:
B-acute lymphoblastic leukaemia (B-ALL) is the most common cancer in children, with 20% of patients relapsing despite major therapeutic advances. A research team of the Development and Genetic Institute in Rennes has identified that the expression of CD9, a transmembrane protein, is linked to the migratory and adhesion capacities of leukaemia cells, enabling them to persist in niches such as the testis. CD9-associated relapses often arise from these niches. Understanding the regulation of CD9 expression is therefore essential.

The hypothesis on which this project is based is that CD9 expression could be orchestrated by ncRNAs. Due to the complexity of deciphering circRNA-miRNA-mRNA networks, an exploration of patient blasts is envisaged in order to delineate a specific non-coding RNA network regulating CD9 expression from bone marrow and blood samples of paediatric-aged patients with B-ALL. If this hypothesis is confirmed, the ncRNAs identified could constitute new specific diagnostic and prognostic markers, or even therapeutic targets.

To confirm this hypothesis, bone and blood sampling of newly diagnosed patients will be collected at the diagnosis, after first phase of treatment and at the relapse, if it occurs.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years
* With established diagnosis of B-ALL
* Initial diagnosis made in the investigating centre
* Having received oral and written information about the protocol, or oral only if the patient is unable to read.
* Having signed a consent form if the patient is capable of giving informed written consent.
* Whose legal guardians have received oral and written information about the protocol, and have signed a free, informed and written consent.
* Beneficiary of a social security scheme

Exclusion Criteria:

* Isolated extramedullary involvement at inclusion
* Patient of childbearing age without effective contraception.
* Adult subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Non coding RNA network in CD9 regulation | 5 years
  description of the network of lncRNAs (circRNAs/miRNAs) involved in the regulation of CD9 present on the surface of blasts at the time of diagnosis of B-ALL (nature of the lncRNAs, level of expression, etc.)

SECONDARY OUTCOMES:
Non coding RNA network in CD9 regulation as a prognosis factor of disease follow-up | 5 years
  Activity of the ncRNA (circRNA/miRNA) network regulating CD9 gene expression as a follow-up marker in CD9+ pediatric B-ALL.
Non coding RNA network in CD9 regulation as a predictive factor of relapse | 5 years
  Activity of the ncRNA (circRNA/miRNA) network regulating CD9 gene expression as a predictive marker of relapse in CD9+ pediatric B-ALL.

CONTACTS AND LOCATIONS:
Overall Officials: Elie COUSIN, Study Chair — Rennes University
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided